CLINICAL TRIAL: NCT06949059
Title: Intravenous Acetaminophen Versus Intravenous Hydromorphone for the Treatment of Acute Pain: A Single-Center, Prospective, Single-Arm Study
Brief Title: Intravenous Hydromorphone for the Treatment of Acute Pain
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Yichang Humanwell Pharmaceutical Co., Ltd., China (Industry)
Responsible Party: Principal Investigator, Hao Sun, Principal Investigator, Clinical Associate Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-320-03
Record Dates: First submitted 2025-04-14; First posted 2025-04-29 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Acute Chest Pain
MeSH Terms: interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): Hydromorphone 1mg was given intravenously and conventional treatment was performed at the same time.
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — Hydromorphone 1mg was given intravenously and conventional treatment was performed at the same time.

SUMMARY:
To observe the efficacy and safety of hydromorphone in the treatment of acute chest pain, and to explore the potential advantages of hydromorphone for analgesia in patients with acute chest pain, so as to provide more theoretical basis for individualized analgesia and rapid recovery in patients with acute chest pain.

ELIGIBILITY:
Inclusion criteria:

1. Age 18-64 years old;
2. Gender is not limited;
3. Patients with acute chest pain, with the time from pain onset to visit the doctor ≤ 24 days;
4. Severe pain that requires the use of opioids to control as determined by emergency physicians;
5. Obtain informed consent from the patient or family members.

Exclusion criteria:

1. Known allergy to hydromorphone or morphine;
2. Systolic blood pressure <100 mmHg, oxygen saturation <95%, pulse less than 60 beats/min;
3. Use of acetaminophen or nonsteroidal anti-inflammatory drugs in the past 8 hours;
4. Chronic pain, defined as pain lasting for more than 12 weeks;
5. Delirium, alcohol withdrawal symptoms or other drug intoxication;
6. Pregnant or lactating women;
7. Patients with mental or neurological diseases, cognitive and consciousness disorders and inability to express correctly;
8. Participating in any other research at the same time;
9. Factors that increase the risk of participating in the study (life-threatening chest pain patients who require rapid diagnosis or treatment intervention, such as resuscitation status, excluding chest pain caused by myocardial infarction), who are judged by the researchers to be unsuitable for inclusion in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Relief at 30 Minutes After Administration | 30 minutes post-medication
  The difference between the NRS pain score before medication and the NRS pain score at 30 minutes after administration (i.e., NRS_before-NRS_at_30min). A larger value indicates a better analgesic effect.

SECONDARY OUTCOMES:
NRS Pain Scores Over 60 Minutes | 0, 5, 15, 30, 45, and 60 minutes after administration (plus 5 minutes after any additional dose)
  NRS pain scores will be measured at baseline (before administration) and at 5, 15, 30, 45, and 60 minutes post-administration. If additional analgesics or rescue medication are given, the NRS is re-measured 5 minutes afterward.
Analgesia Success Rate | Up to 60 minutes post-administration
  The proportion of patients who do not require any additional analgesics within 60 minutes after the initial administration.
Adverse Events Within 60 Minutes | 60 minutes post-administration
  Incidence of adverse events (e.g., hypoventilation, bradycardia, nausea, vomiting, itching, or requirement of naloxone) within 60 minutes after administration.
Total Dose of Rescue Medication | 60 minutes post-administration
  The cumulative dose of any rescue medication administered within 60 minutes after the initial analgesic administration.
Blood Drug Concentration | Baseline; 2, 6, 12, and 24 hours post-administration
  Measurement of drug concentrations from blood samples collected at baseline, 2, 6, 12, and 24 hours after administration, to assess pharmacokinetics.
Oxygen Saturation | Baseline; 15, 30, 45, and 60 minutes post-administration
  Measurement of oxygen saturation recorded at baseline, 15, 30, 45, and 60 minutes post-administration.
Respiratory Rate | Baseline; 15, 30, 45, and 60 minutes post-administration
  Measurement of respiratory rate recorded at baseline, 15, 30, 45, and 60 minutes post-administration.
Systolic Blood Pressure | Baseline; 15, 30, 45, and 60 minutes post-administration
  Measurement of systolic blood pressure recorded at baseline, 15, 30, 45, and 60 minutes post-administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No